CLINICAL TRIAL: NCT01297231
Title: Prospective Analysis of Changes in Background Parenchymal Enhancement (BPE) and Amount of Fibroglandular Tissue on Breast MRI in Early Stage Breast Cancer Patients on Tamoxifen
Brief Title: Prospective Analysis of Changes in Background Parenchymal Enhancement (BPE) and Amount of Fibroglandular Tissue on Breast MRI
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 10-217; Mskcc 10-217 (Other: Memorial Sloan-Kettering Cancer Center)
Record Dates: First submitted 2011-02-14; First posted 2011-02-16 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer
Keywords: fibroglandular tissue; tamoxifen; MRI; Background Parenchymal Enhancement; 10-217
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood or saliva

GROUPS / COHORTS (1):
- Breast cancer: This prospective study will recruit patients with stage 0-3 breast cancer who have had or are scheduled for a breast MRI prior to treatment.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Baseline Breast-MRI within 1 year before starting tamoxifen (allows for surgery, chemotherapy and radiation before the start of tamoxifen).
  During Tamoxifen Treatment:
  * Blood will be drawn for CYP2D6 genotype testing. Analysis of samples will be performed internally at MSKCC.
  * Follow-up breast MRI after 9-12 months of tamoxifen therapy. In patients whom further breast MRI screening and/or follow-up is clinically indicated, follow-up breast MRIs may be performed within 3 months (before or after) the 2, 3, and 4 year time points during tamoxifen treatment. All breast MRIs will be performed using the same technique.
  * Follow-up for all patients during and after tamoxifen should include routine standard clinical assessment and imaging such as mammography and breast MRI when clinically indicated.

SUMMARY:
Tamoxifen is a hormonal treatment for breast cancer. It prevents recurrent disease and decreases death. Tamoxifen is given to women with and at high risk for breast cancer. These women also commonly have breast MRI to monitor for breast cancer. Some features of normal breast tissue visible on breast MRI change depending on patient hormonal status. It has been questioned if hormonal changes due to tamoxifen are seen on breast MRI. Pilot data suggests this is true. If tamoxifen causes changes in normal breast tissue on MRI, more study could be done looking at whether breast MRI could tell us anything about whether tamoxifen is working.

This study is being done to see if tamoxifen changes normal breast tissue on MRI. It will also look at if other factors like taking anti-depressants or gene type have any effect.

ELIGIBILITY:
Inclusion Criteria:

* Females with stage 0-3 breast cancer who have had or are planned to have a breast MRI within 1 year prior to starting tamoxifen
* Premenopausal status is defined as intact ovaries and still menstruating
* Clinical and MRI follow-up planned at MSKCC or MCKCC regional facility
* Willing and able to undergo all study procedures

Exclusion Criteria:

* Contraindication to breast MRI (such as non-compatible cardiac pacemakers or intracranial vascular clips, allergy to Gadolinium)
* Bilateral breast cancer or treatment such as:
* History of or planned bilateral breast irradiation
* History of or planned bilateral mastectomy
* Bilateral breast cancer
* History of unilateral mastectomy or radiation treatment with contralateral breast cancer
* Taking chemo- or hormonal therapy at the time of the baseline breast MRI
* Estrogen and progesterone receptor negative breast cancer
* GFR less than GFR < 30 mL/min/1.73m2
* Postmenopausal women
* Pregnant and/or nursing women
* Less than 21 years of age

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible premenopausal patients with stage 0-3 breast cancer for whom MRI staging is planned will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
To compare the level of BPE on breast MRI | 3 years
  on breast MRI in premenopausal patients with breast cancer before and during 9-12 months on tamoxifen to determine whether tamoxifen results in a significant decrease in BPE and/or amount of fibroglandular tissue

SECONDARY OUTCOMES:
To compare the amount of fibroglandular tissue on breast MRI | 3 years
  on breast MRI in premenopausal patients with breast cancer before and during 9-12 months on tamoxifen to determine whether tamoxifen results in a significant decrease in BPE and/or amount of fibroglandular tissue

CONTACTS AND LOCATIONS:
Overall Officials: Valencia King, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm